CLINICAL TRIAL: NCT05907642
Title: Effects of Dried Plum (Prune) Intake on the Incidence of Low Anterior Resection Syndrome in Patients With Rectal Cancer: a Randomized Controlled Trial.
Brief Title: Effects of Dried Plum (Prune) Intake on the Incidence of Low Anterior Resection Syndrome in Patients With Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ottugi-Prune
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prune (Experimental): During the first 3 days of taking the prunes, 60 g (6 pieces of prune) were consumed per day, and if there were no symptoms corresponding to the safety endpoints for 3 days, the amount was increased to 100 g per day thereafter. Prunes were consumed twice, half each in the morning and afternoon, and the total intake period was 18 days.
  Interventions: Other: Prune (dried plum)
- No-prune (Placebo Comparator): No intervention was provided to the control group, and all normal diets were allowed except for prunes during the study period, for 18 days.
  Interventions: Other: Prune (dried plum)

INTERVENTIONS:
Other: Prune (dried plum) — Subjects who are assigned to the treatment group consume a total of 100 g of prune per day for 18 days and the subjects who are assigned to the control group are allowed to have a normal meal without prune for 18 days.

SUMMARY:
Colorectal cancer is the third leading cause of cancer death and the fourth most commonly diagnosed cancer in the world. The importance of improving the quality of life of patients after colorectal cancer surgery has been gradually emphasized as the survival period after treatment increases. Especially, patients who underwent rectal cancer surgery experience complex bowel movement abnormalities called 'lower anterior resection syndrome' such as urgency, tenesmus, frequent stool passing, which severely degrades the quality of life after surgery. To manage these symptoms, several treatment modalities including medication, neurostimulation, or biofeedback have been tried, but they are not fully effective. Therefore, we designed this clinical trial to examine the effects of dietary supplementation of the fruit, 'Prune', on improving bowel function after anterior resection rectal cancer surgery.

Prune is a dried fruit made from American plums with no seeds, and popular in the worldwide for its sweet and sour flavor and texture. In particular, the high content of sorbitol and dietary fiber softens the stool and improves the overall intestinal function, showing an excellent effect on alleviating constipation symptoms, which has been well studied in several clinical trials.

This study is going to be performed on patients under the age of 65 with primary rectal cancer and rectosigmoid colon cancer who underwent low anterior resection (LAR) exclusive of neoadjuvant chemoradiotherapy. Patients who are treated preoperatively with metallic stent insertion will be excluded. Those who have fruit allergy, diabetes, or chronic constipation will also be excluded. Subjects will be randomly assigned to treatment (Prune) or control group (No-prune) immediately after the surgery. Subjects who are assigned to the treatment group consume a total of 100 g of prune per day and the subjects assigned to the control group are allowed to have a normal meal without prune for 18 days. All subjects should fulfill the LAR syndrome questionnaire, The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-c30), and the defecation habit questionnaire on the day before the surgery and the postoperative day 21. And the subjects also fulfill the defecation diary till the postoperative day 21. The primary endpoint is the incidence of LAR syndrome. The secondary endpoint was the score of EORTC QLQ-C30, defecation habit questionnaire.

Prune intake is less costly than conventional medical treatments for improving bowel function, and it is expected to show high compliance for patients due to the ease of application. Furthermore, if this study demonstrates that prune intake improves the symptoms of LAR syndrome and quality of life after rectal cancer surgery, the ingredients and components of prune could be used to develop new drugs for alleviating the symptoms of LAR syndrome.

ELIGIBILITY:
Inclusion Criteria:

* age 18-69
* tumor located at the rectum or rectosigmoid colon
* who underwent curative surgical resection, low anterior resection

Exclusion Criteria:

* neoadjuvant chemoradiotherapy
* formation of diverting stoma
* preoperative stent insertion
* food allergy
* chronic constipation
* Diabetes mellitus
* previous surgical history of bowel resection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Low Anterior Resection Syndrome Questionnaire Score | Postoperative day 21

SECONDARY OUTCOMES:
The European Organization for Research and Treatment of Cancer quality of life questionnaire c-30 | Postoperative day 21

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No